CLINICAL TRIAL: NCT02184078
Title: An Open-label Study in HIV+ Patients to Determine the Effects of Nevirapine (VIRAMUNE®) on the Steady State Pharmacokinetics of Rifabutin (MYCOBUTIN®)
Brief Title: Study to Determine the Effects of Nevirapine (VIRAMUNE®) on the Steady State Pharmacokinetics of Rifabutin (MYCOBUTIN®) in HIV+ Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1100.1258
Record Dates: First submitted 2014-07-08; First posted 2014-07-09 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Nevirapine; Rifabutin

ARMS (1):
- single group (Experimental): Nevirapine:
  Study days 15-28 dose given once a day (q.d.) Study days 29-42 dose given twice a day (b.i.d.)
  Rifabutin:
  Study Days 0 to 42
  Interventions: Drug: Nevirapine; Drug: Rifabutin

INTERVENTIONS:
Drug: Nevirapine
Drug: Rifabutin

SUMMARY:
Study to determine the effects of nevirapine on the steady state pharmacokinetics of rifabutin and to assess the steady state pharmacokinetics of nevirapine when given in combination with rifabutin

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between the ages of 18 and 65 years who are seropositive for HIV-1 antibody by an ELISA test and confirmed by an alternative method e.g. Western Blot
* Lymphocytes Expressing CD4+ Surface Marker (CD4+ cell count) >= 100 cells/mm³
* Patients must be taking at least 2 antiretroviral agents (with the exception of ritonavir, nelfinavir and non-nucleoside reverse transcriptase inhibitors taken continuously for at least 28 days prior to study entry (Day 0)
* Patients currently being treated with rifabutin during the screening period may be included provided that patients are receiving 300 mg once daily (or 150 mg once daily for patients concomitantly taking Zidovudine (ZDV), saquinavir or indinavir) and that there has been no change in dosing of > 25% within 28 days prior to Study Day 0
* Patients who meet the following laboratory parameter:

  * Granulocyte count > 1000 cells/mm³
  * Hemoglobin > 9.0 g/dl (men and women)
  * Platelet count > 75000 cells/mm3
  * Alkaline Phosphatase < 3.0 times the upper limit of normal
  * Serum Glutamic-Oxaloacetic Transaminase (SGOT) and Serum Glutamic-Pyruvic Transaminase (SGPT) < 3.0 times the upper limit of normal
  * Total bilirubin < 1.5 times the upper limit of normal
* Female patients of childbearing potential must be willing to use a reliable form of contraception which must include a medically form of barrier contraception
* Patients able to provide written consent and comply with study requirements

Exclusion Criteria:

* Female patients who are pregnant or breast-feeding
* Seated systolic blood pressure below 100 mmHg or greater than 150 mmHg and/or heart rate less than 50 or greater than 90 beats/min.
* History of drug allergy or known drug hypersensitivity
* Patients receiving any investigational drug, antineoplastic agent or radiotherapy other than local skin radiotherapy treatment within 12 weeks before starting study medication
* Patients requiring systemic treatment with corticosteroids or drugs known to be hepatic enzyme inducers or inhibitors within 14 days of study entry (Study Day 0). Such substances in theses categories include: macrolide antibiotics (erythromycin, clarithromycin, azithromycin) azole antifungals (ketoconazole, fluconazole, itraconazole) rifampin and phenytoin
* Use of ritonavir, nelfinavir or non-nucleoside reverse transcriptase inhibitors within 28 days of Study Day 0 or during the trial
* Patients with clinical evidence of active tuberculosis (TB) or undergoing treatment or prophylaxis for TB
* Patients with a current history of intravenous drug abuse, alcohol or substance abuse (within the last year)
* History of any clinically important disease including hepatic, renal, cardiovascular or gastrointestinal
* Patients with malabsorption, severe chronic diarrhea or subject unable to maintain adequate oral intake
* Patients with no previous antiretroviral background therapy taken continuously for the 28 days prior to study entry (Day 0)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 1998-10; Primary Completion 1998-12 (Actual)

PRIMARY OUTCOMES:
Cmax,ss (maximum observed concentration at steady state) | predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post dose at day 14 and day 42
Cmin,ss (minimum observed concentration at steady state) | predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post dose at day 14 and day 42
Tmax,ss (Time of Cmax at steady state) | predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post dose at day 14 and day 42
Area under the plasma concentration time curve over the dosing interval | predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post dose at day 14 and day 42
CL/F (apparent total clearance) | predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post dose at day 14 and day 42

SECONDARY OUTCOMES:
Number of patient with adverse events | up to day 43